CLINICAL TRIAL: NCT03063684
Title: Fractional / Pixel CO2 Laser Treatment of Vulvar Atrophy and Lichen Sclerosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Ahinoam Lev-Sagie, MD, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0598-16-HMO
Record Dates: First submitted 2017-02-18; First posted 2017-02-24 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Vaginal Atrophy; Lichen Sclerosus
MeSH Terms: conditions — Lichen Sclerosus et Atrophicus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaginal atrophy (Experimental): With decreasing estrogen levels occurring following menopause, changes of the vaginal mucosa appear: it becomes thin and pale and loses its elasticity. The blood supply decreases, normal secretion is reduced, the epithelial cells do not undergo the normal differentiation process, the bacterial population changes with loss of lactobacilli and pH increases. These changes are associated with morphological and histological changes, manifested, among other findings, by alterations in the collagen composition, loss of the trabecular organization of collagen and reduced amount of elastic fibers. Women with reduced vaginal estrogen content may report dryness, itching, discomfort, burning sensation during micturition, pain and dyspareunia. These changes are reversible: topical or systemic estrogen change the vaginal mucosa's characteristics and may also alleviate complaints arising from estrogen deficiency.
  The intervention is 3 treatments with fractional / Pixel CO2 Laser
  Interventions: Device: Fractional / Pixel CO2 Laser
- Lichen sclerosus (Experimental): Lichen sclerosus is a chronic cutaneous disease involving the vulvar and peri-anal skin. The involved skin becomes thin and white, with frequently present bruises or petechiae and anatomic changes.
  Lichen sclerosus is thought to be an auto-immune disorder and its most frequent signs are itching, irritation or burning. The discoloration may involve the entire vulvar and peri-anal area (sometimes having the form of an "8" or a "keyhole" surrounding the vulva and anus) or appear as separated spots of various sizes occupying only part of the skin. At advanced stages of lichen sclerosus, scarring may appear, with loss of the labia minor and adhesions which may entirely cover the clitoris.
  The treatment is of topical steroid. Lichen sclerosus is a chronic disorder, and even with good treatment, in a certain proportion of cases the skin does not return to its original appearance.
  The intervention is 3 treatments with fractional / Pixel CO2 Laser
  Interventions: Device: Fractional / Pixel CO2 Laser

INTERVENTIONS:
Device: Fractional / Pixel CO2 Laser — The laser energy is transferred in a fractioned manner: the laser beam splits while passing through a lens to 81 dots (9 x 9 pixels) onto approximately 1 cm2, so the laser rays hit the tissue in small spots.
  For gynecological applications, the treatment is performed by a transducer, which was specifically designed for vaginal application.

SUMMARY:
The study will examine the effects of fractional/pixel CO2 laser treatment in vaginal atrophy and in vulvar lichen sclerosus by means of histological and immuno-histochemical characterization of the epithelial layers and markers of tissue aging. The tissue characterization will be performed by biopsies of the vaginal or vulvar tissue at three different points of time: prior to treatment, two weeks after the third and last treatment, and one year after the last treatment.

DETAILED DESCRIPTION:
Many studies have been published recently describing the use of a fractional/pixel CO2 laser for the treatment of various disorders of the vulva and the vagina, such as atrophy due to estrogen deficiency, urinary stress incontinence, skin diseases (lichen sclerosus) and more.

The results of the studies that investigated this technology in relation to vaginal atrophy and urinary stress incontinence have shown improvement in symptoms after a series of only 3 treatments.

The proposed effect of the fractional CO2 laser is based on studies performed on non-genital tissues [Daffon, Capon], which demonstrated changes in the connective tissue and proliferation of fibroblasts, as well as formation of collagen and elastic fibers. The suggested explanation is based on the theory that heat shock proteins are involved in the process and arise due to thermal tissue damage, and this in turn activate tissue cytokines, growth factors and fibroblasts. These theories have not been proven for vulvar and vaginal tissues, and except for the demonstration of histologic and morphologic changes in the irradiated tissues [Salvatore, Menopause 2015], the cellular mechanism of action and the nature of the process mediating the changes in uro-genital tissues has not yet been examined.

The technology known as fractional CO2 has been used for many years in dermatology and plastic surgery. In this method, the laser beam splits while passing through a lens to 81 dots (9 x 9 pixels) onto approximately 1 cm2. The laser beam penetrates the tissue and causes minimal evaporation around each spot of the fractionated beams and release of heat only at the desired tissue depth. The method of energy transfer to tissues in tiny dots leads to the creation of various thermal effects in the focus of the beam, around the focus, and in the areas between these heat foci. Following the tissue irradiation, different processes occur: epithelial cell proliferation and thickening of the epithelial layer, migration and proliferation of endothelial cells, creation of neo-vasculature in the lamina propria, creation of collagen and elastic fibers, and accumulation of glycogen in the cells [Salvatore, Menopause 2015]. The result of these processes is improved tissue elasticity and plasticity as well as regeneration of the epidermis layer. Previous studies demonstrated that the effect of this treatment on the atrophic vagina is identical to long-term local estrogen treatment, with improved cytological index, improved lubrication, alteration of the vaginal flora, and reduced acidity to the level of "estrogenic" levels (approx. pH 4 -4.5) [Salvatore, Menopause, 2015;Perino; Gasper; Salvatore, Climacteric, 2015].

Considering the multitude of recently published articles presenting impressive clinical results, the investigators decided to examine the effects of the treatment with a fractional CO2 laser on the vaginal and vulvar tissue at a cellular level for two conditions: vaginal atrophy due to estrogen deficiency and lichen sclerosus. These two conditions were chosen due to the magnitude of recent publications dealing with clinical and histological improvement in these two pathological conditions following laser treatment. Understanding the cytological processes will enable the foundation of knowledge about the basic mechanism of action, and propose methods to improve the current therapeutic protocols. It will also enable the observation of the duration of the treatment effect, and the assessment of whether these changes are associated with undesired events, such as increased risk of malignant tissue transformation.

Patients The investigators intend to recruit 10 women for each group (10 women with atrophy and 10 with lichen sclerosus). Considering the availability of efficient and safe medical treatment, most women diagnosed with lichen sclerosus or vaginal atrophy are treated with medical preparations to their satisfaction. Therefore, the investigators will recruit the following types of patients for the trial: women with low compliance for the medical treatment, women who have developed intolerance to the treatment (such as chronic candida vulvovaginitis under long-term estrogen treatment, hypersensitivity reactions to the steroid ointment or estrogen preparation, or drug allergy) or women with only partial response to treatment, for whom there is no satisfactory therapeutic alternative.

The study includes 6 appointments:

T0-recruitment: ascertain eligibility, sign informed consent form, complete a questionnaire including epidemiologic and clinical details, gynecological examination, cytological smear (maturation index), determination of the acidity level of the vaginal secretions (pH), determination of vaginal health index score [Bachmann].

A punch biopsy will be taken from the mid-third of the vagina (in vaginal atrophy) or the vulva (in lichen sclerosus).

T1-Visit 2 (2-4 weeks from recruitment) The treatment protocol includes a series of three laser treatments, 4-6 weeks apart.

The first laser treatment will be performed during Visit 2. In the vagina, the treatment is performed by a special vaginal transducer enabling 360° treatment; the irradiation of the vagina is performed in adjacent "squares" along the entire vaginal circumference, by turning the handle while slowly withdrawing the transducer from the vaginal canal. The duration of treatment is 5-7 minutes. The vaginal treatment is not associated with pain. The treatment of the introitus will be performed by a transducer enabling treatment around 360° named FemiLift.

The treatment will be performed by a fractional micro-ablative CO2 laser system manufactured by Alma Laser in accordance with the accepted protocol (laser mode: pulse, energy: 40-80 mj/pulse).

For lichen sclerosus, a handgrip of the FemiLift transducer will be used, which transmits the "pixel print" directly and not under a 90° angle. Since the vulvar skin is pain sensitive, it will be treated prior to the laser application, with EMLA anesthetic cream. The duration of treatment is 3-7 minutes and it is performed by the same device with energy levels of 20-60 mj/pulse.

During Visit 3 (T2) and Visit 4 (T3), identical treatment to that described above will be performed.

In the framework of the study, the below follow-up procedures will be performed:

1. Biopsy - three biopsies will be taken from the lateral mid-third of the vagina: prior to treatment (T0), two weeks after the third and final treatment (T4) and one year after the completion of the treatment series (T5). The biopsy will be a punch biopsy with a 5 mm diameter. The biopsies will be performed under local anesthesia with 2% lidocaine.
2. In the course of each of the follow-up examinations (T 0 - 5), the following will be performed (In vaginal atrophy):

   * Gynecological examination with speculum
   * Smear taken from the mid-third of the vagina with a cotton tip applicator, which will be used for a cytological smear and to determine the acidity level of the vaginal secretions.
   * The vaginal health index score will be determined, including the evaluation of 5 parameters: elasticity, pH, integrity of the epithelium, moisture and fluid volume. Each parameter is scored on a scale of 1 to 5, and if the total score is lower than 15, the vagina is considered atrophic [Bachmann].
   * The patient will be requested to grade symptoms (dryness, itching, burning, discomfort, dyspareunia, dysuria) on a VAS (visual analog scale) with "very disturbing" and "not disturbing at all" at its limits.
   * The patient will be requested to grade the extent of her satisfaction with the treatment results (very satisfied. satisfied, not sure, not satisfied, very unsatisfied).
   * The patient will be requested to report side effects.

In lichen sclerosus patients:

- External examination of the vulva and a photograph of the results for follow-up.

The biopsies will be sent to the Institute of Pathology at Hadassah Hospital, where the following examinations will be performed:

1. Routine hematoxylin-eosin staining.
2. Immunohistochemistry staining for P16 protein.
3. Immunohistochemistry staining for the KI-67 protein.
4. Immunohistochemistry staining for the p63 protein,\.
5. Staining for alpha and beta estrogen receptors and progesterone receptors.

ELIGIBILITY:
Vaginal Atrophy - Inclusion Criteria

* Menopause for more than one year
* One or more of the following symptoms: sensation of dryness, itch, irritation, burning, discomfort, dysuria, dyspareunia
* Characteristic atrophic changes on gynecological examination
* Laboratory workup: pH >4.5, characteristic microscopic smear (increased number of para-basal cells)
* Normal Pap-smear within 12 months
* Negative vaginal culture for fungi or relevant bacteria
* Negative test for STD pathogens (chlamydia, gonorrhea, genital mycoplasma and trichomonas)

Exclusion Criteria

* Genital skin disease
* Active infection
* Pelvic organs prolapse above grade 2
* Previous surgery for pelvic organs prolapse
* Use of systemic or local hormonal preparations during 6 months preceding the study treatment
* History of malignant diseases
* Undiagnosed vaginal bleeding
* Use of analgesics or antidepressants
* Use of anticoagulants

Lichen Sclerosus Inclusion Criteria

* Age 18-80
* Biopsy demonstrates characteristic changes for lichen sclerosus
* One or more of the following symptoms: sensation of dryness, itch, irritation, burning, discomfort.
* Characteristic changes for lichen sclerosus on gynecological examination
* Negative vaginal culture for fungi or relevant bacteria
* Negative test for STD pathogens (chlamydia, gonorrhea, genital mycoplasma and trichomonas)

Exclusion Criteria

* Use of steroid-containing creams for the vulvar region two months preceding recruitment
* Additional genital skin disease
* Active infection
* History of malignant diseases
* Use of analgesics or antidepressants
* Use of anticoagulants
* Pregnancy or planning pregnancy during the study
* Systemic treatment with immuno-modulatory drugs

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-04-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline of vaginal health index score | T0-Recruitment, T1-2-4 weeks, T2- 6-8 weeks, T3-10-12 weeks, T4-12-14 weeks, T5- 12 months
  Score of 1-15, which includes the following parameters: elasticity, fluid volume, pH, epithelial integrity, moisture.

SECONDARY OUTCOMES:
Change from baseline of Maturation Index | T0-Recruitment, T1-2-4 weeks, T2- 6-8 weeks, T3-10-12 weeks, T4-12-14 weeks, T5- 12 months
  Ratio of parabasal cells, intermediate cells and mature squamous cells
Change from baseline of pH measurement | T0-Recruitment, T1-2-4 weeks, T2- 6-8 weeks, T3-10-12 weeks, T4-12-14 weeks, T5- 12 months
Change from baseline of patient's symptoms | T0-Recruitment, T1-2-4 weeks, T2- 6-8 weeks, T3-10-12 weeks, T4-12-14 weeks, T5- 12 months
  Visual analogue scale of symptoms (dryness, itch, irritation, pain, dysuria and dyspareunia)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dafforn TR, Della M, Miller AD. The molecular interactions of heat shock protein 47 (Hsp47) and their implications for collagen biosynthesis. J Biol Chem. 2001 Dec 28;276(52):49310-9. doi: 10.1074/jbc.M108896200. Epub 2001 Oct 9. PMID 11592970
- [Background] Capon A, Mordon S. Can thermal lasers promote skin wound healing? Am J Clin Dermatol. 2003;4(1):1-12. doi: 10.2165/00128071-200304010-00001. PMID 12477368
- [Background] Salvatore S, Leone Roberti Maggiore U, Athanasiou S, Origoni M, Candiani M, Calligaro A, Zerbinati N. Histological study on the effects of microablative fractional CO2 laser on atrophic vaginal tissue: an ex vivo study. Menopause. 2015 Aug;22(8):845-9. doi: 10.1097/GME.0000000000000401. PMID 25608269
- [Background] Perino A, Calligaro A, Forlani F, Tiberio C, Cucinella G, Svelato A, Saitta S, Calagna G. Vulvo-vaginal atrophy: a new treatment modality using thermo-ablative fractional CO2 laser. Maturitas. 2015 Mar;80(3):296-301. doi: 10.1016/j.maturitas.2014.12.006. Epub 2014 Dec 25. PMID 25596815
- [Background] Gaspar A, Brandi H, Gomez V, Luque D. Efficacy of Erbium:YAG laser treatment compared to topical estriol treatment for symptoms of genitourinary syndrome of menopause. Lasers Surg Med. 2017 Feb;49(2):160-168. doi: 10.1002/lsm.22569. Epub 2016 Aug 22. PMID 27546524
- [Background] Salvatore S, Nappi RE, Parma M, Chionna R, Lagona F, Zerbinati N, Ferrero S, Origoni M, Candiani M, Leone Roberti Maggiore U. Sexual function after fractional microablative CO(2) laser in women with vulvovaginal atrophy. Climacteric. 2015 Apr;18(2):219-25. doi: 10.3109/13697137.2014.975197. Epub 2014 Dec 16. PMID 25333211
- [Background] Bachmann GA, Notelovitz M, Kelly SJ, et al: Long-term nonhormonal treatment of vaginal dryness. Clin Pract Sex 8:8, 1992